CLINICAL TRIAL: NCT06686173
Title: The Effect of the Parous Female and Young Male Donor on the Outcomes of GVHD Prophylaxis Underwent the Combined Treatment of ATG and PTCy for Haplo-HSCT: a Prospective, Multi-center, Cohort Study
Brief Title: Effect of Donor Chose on the Outcomes of GVHD Prophylaxis Underwent the Combined Treatment of ATG/PTCy for Haplo-HSCT
Acronym: Donor chose
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, professor of medicine, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: SHSYXY-haplo-PBSCT-donor
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: High-Risk Acute Myeloid Leukemia; Relapse And/or Refractory AML
MeSH Terms: interventions — Donor Selection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — the bone marrow and peripheral Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: None-placebo — This is one kind descriptive study. The different donor groups made the cohorts different: the parous female donor and young male donor
Other: non-intervention study — This study is one kind of non intervention study
Other: donor selection — the intervention of this study was the different donor groups: the parous female donor and young male donor. All the patients involved in this study were treated by the combination of ATG and PTCy

SUMMARY:
This is a prospective, multicenter, cohort study. The high-risk, relapse and refractory AML patients were enrolled in this study. And the goal of this study is to study the effect of the parous female donor and young male donor on the outcomes of graft-versus-host disease (GVHD) prophylaxis underwent the combination of ATG and PTCy for haploidentical peripheral blood stem cell transplantation

ELIGIBILITY:
Inclusion Criteria:

1. Acute myeloid leukemia was diagnosed according to the 2016ELN criteria with any of the following:

1. ELN prognostic stratification high-risk group (see Appendix for criteria)
2. Non-remission (NR) AML: including primary refractory AML and NR patients after relapse.

2. Patients must have a suitable hematopoietic stem-cell donor.

1. Patients had to have a qualified haploidentical young male (≤30 years old) or female with a history of pregnancy;
2. Related donors had to be related donors matched 5/10-7/10 for HLA-A, -B, -C, -DQB1 and -DRB1 3. All the enrolled patients received a unified GVHD prevention regimen based on ATG and PTCy

Exclusion Criteria:

1. Intermediate-low risk AML patients (ELN criteria);
2. Patients with extramedullary active lesions at the time of transplantation;
3. Haploidentical collateral donors;
4. Patients who refused allogeneic hematopoietic stem cell transplantation;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The high-risk, relapse and refractory AML patients were enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
RFS | one year
  1-year RFS after transplantation